CLINICAL TRIAL: NCT05129449
Title: Safety and Performance of the Motorized Spiral Endoscope PowerSpiral in Subjects Indicated for Small-bowel Enteroscopy or Endoscopic Retrograde Cholangio-Pancreatography (ERCP) in Subjects With Surgically Altered Gastrointestinal Anatomy.
Brief Title: A Clinical Study With the Medical Device PowerSpiral for Endoscopic Retrograde Cholangio-Pancreatography (ERCP)
Acronym: SAMISEN-B
Status: Completed | Type: Observational
Sponsor: Olympus Europe SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-GI (OEKG) - 01 Phase B
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-07

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endoscopic Retrograde Cholangio-Pancreatography (ERCP) — Endoscopic Retrograde Cholangio-Pancreatography (ERCP) conducted with motorized PowerSpiral in subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication.

SUMMARY:
The objective of the SAMISEN study phase B is to assess the performance and safety of diagnostic and therapeutic procedures with the Olympus Motorized Spiral Enteroscope (PowerSpiral) in subjects with surgically altered gastrointestinal anatomy indicated for an Endoscopic Retrograde Cholangio-Pancreatography (ERCP).

DETAILED DESCRIPTION:
The main objective of this registry is to collect data on the safety and performance of the motorized PowerSpiral device during Post-market Clinical Follow-up in subjects with surgically altered gastrointestinal anatomy indicated for an Endoscopic Retrograde Cholangio-Pancreatography (ERCP). It is assumed that this motorized PowerSpiral device and its safety profile is non-inferior to preceding generations of balloon assisted enteroscopes.

As clinical performance and efficacy is equally important for the user this study also collects efficacy and handling data of the motorized PowerSpiral device.

ELIGIBILITY:
Inclusion criteria

1. Signed informed consent
2. Patients with surgically altered upper Gastrointestinal anatomy (Roux-en-Y and Billroth II types) with a biliary indication for ERCP where access with conventional ERCP devices is of no avail and after careful risk assessment.

Exclusion criteria In addition to be eligible for study enrollment a subject must not meet any of the exclusion criteria listed below.

1. Age under 18 years
2. Female and of child-bearing age who is currently pregnant or planning to become pregnant within the study period
3. Any contraindication to standard enteroscopy or ERCP (e.g. severe coagulopathy or known coagulation disorder; bowel obstruction / stenosis, stents or other instruments implanted in the intestinal tract, suspected GI perforation, esophageal or gastric varices, eosinophilic esophagitis) as judged by the investigator after careful individual risk assessment
4. Concurrent participation in another competing clinical study
5. Pancreatic indication for ERCP in patient with surgically altered anatomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication, which fulfil all inclusion and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Beyna, MD PhD, Principal Investigator — Evangelisches Kranken-haus Düssel-dorf; Tom G. Moreels, Prof., Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (5):
- Belgium (2):
  - Cliniques universitaires Saint-Luc, Brussels
  - Hôpital Erasme, Brussels
- Germany (2):
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - University Hospital Frankfurt a.M., Frankfurt
- OUS-Rikshospitalet University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreels TG, Aabakken L, Arvanitaki M, Knabe M, Beyna T. Enteroscopy-assisted ERCP in patients with surgically altered anatomy: Multicenter prospective registry (SAMISEN-B) using motorized spiral enteroscopy. Endosc Int Open. 2024 Nov 28;12(11):E1392-E1400. doi: 10.1055/a-2443-1514. eCollection 2024 Nov. PMID 39610946

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Study: All patients received an ERCP examining with the CE- marked PowerSpiral (OLYMPUS PSF-1, SINGLE USE POWER SPIRAL TUBE and motor control unit POWER SPIRAL CONTROL) device.
Period: Overall Study
Arm/Group | Single Arm Study
Started | 89
Completed | 88
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study
Number analyzed (Participants) | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (15.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 35
  Norway | 13
  Germany | 40

OUTCOME MEASURES:

1. Primary Outcome: Total Success Rate. Defined as the Combined Percentage of Enteroscopy Success Rate, Biliary Cannulation Success Rate and Procedural (Therapeutic) Success Rate.
Description: The total success rate refer to the percentage of the following succes rates relevant for ERCP procedures. Combined percentage of Enteroscopy success rate, Biliary Cannulation success rate and Procedural (Therapeutic) success rate.
Time Frame: 17 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 88
Participants | 45

2. Primary Outcome: Total Procedure Time
Description: starting with oral insertion until final withdrawal of the device
Time Frame: Same day of the ERCP measurement.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Single Arm Study
Number analyzed (Participants) | 88
Minutes | 71.1 (42.4)

3. Primary Outcome: Enteroscopy Time
Description: starting with oral insertion until reaching the papilla or the biliary anastomosis
Time Frame: Same day of the ERCP measurement.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Single Arm Study
Number analyzed (Participants) | 88
Minutes | 29.4 (22)

4. Primary Outcome: (Serious) Adverse Events and Device Deficiencies.
Description: Incidence (% of subjects) and frequency (no. of subjects) with Serious Adverse Events (SAEs) and Device Deficiencies (DD) which meet the severity grading of moderate or severe for the following categories:
  * Enteroscopy-associated complications (mainly bleeding and perforation(s))
  * ERCP-related complications (Dumonceau et al. 2020)
  * Sedation / anesthesia related complications
  * other
Time Frame: 17 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 88
Participants
  Serious Adverse Events (SAE) | 6
  Device deficiency | 1
  None SAE and devive deficiency | 81

ADVERSE EVENTS:
Time Frame: 17 months
Arm/Group | Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/88
Serious Adverse Events (participants affected / at risk) | 6/88
Other Adverse Events (participants affected / at risk) | 6/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=88)
Bleeding (Gastrointestinal disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2)
Perforation (Gastrointestinal disorders) | 2 (2)
Suspected pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=88)
Bleeding (Gastrointestinal disorders) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Other (System malfunction, non-rotation of spiral before start.) (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT05129449/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT05129449/SAP_001.pdf